CLINICAL TRIAL: NCT04400669
Title: The Effect of Mechanical Bowel Preparation Prior to Gynaecological Laparoscopic Surgeries on the Pressure of Pneumoperitoneum and Trendelenburg Inclination Angle During the Surgery: A Novel Perspective for Patient Safety
Brief Title: The Effect of Mechanical Bowel Preparation Prior to Gynaecological Laparoscopic Surgeries on the Surgical Conditions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Kadir Bakay, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MBP
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Patient Preference; Patient Safety
Keywords: mechanical bowel preparation; gynecological surgery; Minimally invasive gynecological procedures; Enema; Trendelenburg angle; Pneumoperitoneum pressure
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Surgeons and the assessor will be blind. The nurse working in the gynecology setting perform the intervention to the previously randomized patients. Patient will be told for not to reveal the intervention that she undergoes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mechanical Bowel Preparation (Experimental): Patients will have only clear liquids after a normal breakfast and lunch on the day before surgery and subsequently fasten for 7-9 hours prior to surgery. Patients will ingest first dose of 45 ml oral sodium phosphate (NaP) enema (BT ORAL SOLUSYON 45 ML®, Yenisehir Lab. Tic. San. Ltd. Sti, Turkey) at 4 p.m. and a second dose at 8 p.m. in the evening before the scheduled surgery.
  Interventions: Other: Mechanical Bowel Preparation
- Low fibre diet (Active Comparator): Patients will be given detailed instructions about the pre-operative diet (total daily Fibre intake inferior to 10 g) to be used for 3 days prior to surgery.
  Interventions: Dietary Supplement: Low fibre diet
- MBP plus low fibre diet (Active Comparator): This group will receive both mechanical bowel preparation and 3-days low fibre diet.
  Interventions: Other: MBP plus low-fibre diet
- Control (No Intervention): Control subjects will receive no instructions about the pre-operative diet (free diet).

INTERVENTIONS:
Other: Mechanical Bowel Preparation — oral sodium phosphate (NaP) enema
  Arms: Mechanical Bowel Preparation
Dietary Supplement: Low fibre diet — 3 days
  Arms: Low fibre diet
Other: MBP plus low-fibre diet — 3 days low fibre diet preoperative mechanical bowel preparation
  Arms: MBP plus low fibre diet

SUMMARY:
This RCT aims to investigate the real surgical effects of MBP prior to the gynecological laparoscopic surgeries. Those effects include lowest pneumoperitoneum pressure, lowest Trendelenburg inclination angle, the ease of the surgical view and the preferences of the patients with objective measures.

DETAILED DESCRIPTION:
Mechanical bowel preparation (MBP) has been routinely used prior to minimally invasive gynaecologic procedures (MIGP) hypothetically to improve intraoperative bowel handling and visualization of the surgical field, and also to reduce faecal contamination in the setting of bowel injury and/or resection.

The studies investigating the effect of MBP on MIGP are limited and most of existing data are extrapolated from the reports of colorectal and urological surgery studies.

Besides, evaluation of the surgical workspace visualization and intraoperative bowel handling are far from being objective since they were mostly measured by a 4/5/10-point Likert scales or rated verbally on scales of excellent to poor by the operating surgeons.

In contrary, it is planned to use objective visualize index, and objective surgical conditions to measure whether MBP has any effect or not.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Able to provide informed consent
* Undergo laparoscopic gynecological surgery for a benign condition

Exclusion Criteria:

* History of previous abdominal surgery
* Clinically significant present or past systemic diseases
* Inability to perform mechanical bowel preparation
* Suspicion of malignancy
* Association with non-gynaecological surgical pathologies
* Severe endometriosis (stage ≥ III according to the classification of the American Society for Reproductive Medicine)
* Psychiatric disorders precluding consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-11-05 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
The surgical visibility of abdomen | After the introduce of first left lateral port
  A scale title as "Objective Visual Indexing (OVI)" will be used for assessing the visibility of the Douglas pouch and adnexa. The assessment of the visibility of Douglas pouch and adnexa will be performed under standard pneumoperitoneum pressure (12mmHg) and Trendelenburg inclincation angle (30). After the first Inspection, scale of VI scoring will be calculated by adding up the points obtained from optical inspection. Higher scores mean better visuality of the surgical field.
The lowest pneumoperitoneum pressure (PP) at standard Trendelenburg inclination angle (TIA). | In the initial phase of the surgery
  The PP will be increased to 15 mmHg while keeping the TIA same, at 30o. The surgeon will displace the bowel beginning from the cecum followed by the last ileal loop above the sacral promontory. Once the bowel was displaced out of the pelvis, the PP will be stepwise decreased by 1 mmHg during 1 min intervals to the lowest pressure where the bowel is to descend towards the pelvis over the pelvic brim and/or where the surgical workspace is not adequate to proceed safely with the planned operation. This value will be recorded as the lowest PP adequate to proceed safely with the planned surgery at standard TIA (30 degree).
The lowest Trendelenburg inclination angle (TIA) at standard pneumoperitoneum pressure (PP) adequate to proceed with the planned operation. | In the initial phase of the surgery
  The PP obtained in outcome 2 will be readjusted to the standard 12 mmHg keeping the TIA same, at 300. Then, the surgeon will replace the bowel beginning from the cecum followed by the last ileal loop above the sacral promontory. Once the bowel is displaced out of the pelvis, the TIA will be gradually decreased by 1o with 15 seconds intervals to the degree where the bowel is to descend towards the pelvis over the pelvic brim. This value will be recorded as the lowest TIA adequate to proceed safely with the planned surgery at standard PP (12 mmHg).

SECONDARY OUTCOMES:
Preoperative patient symptomatology | Right before the surgery
  Patients will be interviewed in the preoperative holding area or in the patient's room about the acceptability of the intervention (MBP / diet) and adverse pre-operative events, including: nausea, insomnia, headache, thirst, weakness, tiredness, discomfort, abdominal cramps, sleep disturbances. These symptoms will be scored with using a 10-cm "Visual Analog Score" (VAS). Higher scores mean worse outcome.
Postoperative pain | at 24th hours
  The intensity of the postoperative pain was measured by an independent investigator at 24th hours with a 10-cm Visual Analog Score (VAS). Higher scores mean worse outcome.
Complications | At 1st week and 6th week postoperatively or whenever it occurred.
  Intraoperative complications, at 1st week and 6th week postoperatively, between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kadir Bakay, Assoc Prof, Principal Investigator — Ondokuz Mayis Universitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Egemed Hospital, Aydin
  - Samsun Medical Faculty, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Raw data (for meta-analysis), statistical analyses and study protocol can be shared upon request. Processed data can be shared after completion of the study.
Supporting Information: Study Protocol, CSR
Time Frame: After the completion of the study, for 10 years.
Access Criteria: Access will be granted right after establishing a contact.
URL: https://drive.google.com/file/d/1E5qV7Ff_ltsXFYc0m4MgO2a4N-BmVRSQ/view?usp=sharing

REFERENCES:
- [Result] Bakay K, Aytekin F. Mechanical bowel preparation for laparoscopic hysterectomy, is it really necessary? J Obstet Gynaecol. 2017 Nov;37(8):1032-1035. doi: 10.1080/01443615.2017.1318268. Epub 2017 Jun 26. PMID 28650683